CLINICAL TRIAL: NCT03760731
Title: Thriving in the Midst of Moral Pain: The Acceptability and Feasibility of Acceptance and Commitment Therapy for Moral Injury (ACT-MI) Among Warzone Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA Palo Alto Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D2854-R; 1I01RX002854-01A1 (NIH)
Record Dates: First submitted 2018-11-29; First posted 2018-11-30 (Actual); Results first posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Moral Injury
Keywords: Psychosocial Rehabilitation; Acceptance and Commitment Therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Acceptance and Commitment Therapy for Moral Injury (ACT-MI) is a novel treatment protocol detailing the application of ACT to help Veterans learn to interact differently with moral emotions and engage meaningfully in their lives. The intervention is group-based and spans fifteen weeks and is a hybrid of twelve, 90-minute psychotherapy group sessions and three, 30-minute individual case conceptualizing sessions. The current ACT-MI protocol was developed through an iterative process in which authors generated and refined the intervention based on clinical interactions with Veterans currently reporting moral injury.
  Present Centered Therapy for Moral Injury (PCT-MI) represents a 15-week protocol consisting of twelve 90-minute group sessions and three 30-minute individual case conceptualizing sessions, but will focus on problem solving daily life difficulties related to moral injury rather than the experiential focus on moral emotions presented in ACT-MI.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will be blind to treatment condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acceptance and Commitment Therapy for Moral Injury (ACT-MI) (Experimental): Acceptance and Commitment Therapy for Moral Injury (ACT-MI) is a novel treatment protocol detailing the application of ACT for recovery from moral injury. ACT-MI is designed to help Veterans learn to interact differently with moral emotions and engage meaningfully in their lives. The intervention is group-based and spans fifteen weeks including 12, 90-minute group sessions and 3, 30-minute individual case conceptualizing sessions. The current ACT-MI protocol was developed through an iterative process in which authors generated and refined the intervention based on clinical interactions with Veterans currently reporting moral injury.
  Interventions: Behavioral: Acceptance and Commitment Therapy for Moral Injury (ACT-MI)
- Present Centered Therapy for Moral Injury (PCT-MI) (Active Comparator): Present Centered Therapy (PCT-MI) represents a 15-week intervention with 12 90-minute group sessions and 3 30-minute individual case conceptualizing sessions. PCT-MI focuses on problem solving daily life difficulties related to moral injury rather than the experiential focus on moral emotions presented in ACT-MI. Because PCT has been established as an evidence-based active control condition, it is likely to serve as a beneficial transdiagnostic intervention in its own right. PCT-MI could provide another treatment option that might be preferable to some Veterans and promote patient choice. Additionally, PCT-MI would require less clinician training and specialization than ACT-MI. Using PCT-MI as an active comparison condition will determine whether it is necessary to train clinicians in ACT-MI or if therapists with exposure to supportive problem-solving therapy approaches can lead a group that impacts functioning among Veterans reporting moral injury-related distress.
  Interventions: Behavioral: Present Centered Therapy for Moral Injury (PCT-MI)

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy for Moral Injury (ACT-MI) — Acceptance and Commitment Therapy for Moral Injury (ACT-MI) is a novel treatment protocol detailing the application of ACT for recovery from moral injury. ACT-MI is designed to help Veterans learn to interact differently with moral emotions and engage meaningfully in their lives. The 15-week intervention spans twelve, 90-minute group sessions and 3 30-minute individual case conceptualizing sessions. The current ACT-MI protocol was developed through an iterative process in which authors generated and refined the intervention based on clinical interactions with Veterans currently reporting moral injury.
  Other Names: ACT-MI
  Arms: Acceptance and Commitment Therapy for Moral Injury (ACT-MI)
Behavioral: Present Centered Therapy for Moral Injury (PCT-MI) — Present Centered Therapy for Moral Injury (PCT-MI) is a 15-week intervention consisting of 12 90-minute group sessions and 3 30-minute individual case conceptualizing sessions, focused on problem solving daily life difficulties related to moral injury rather than the experiential focus on moral emotions presented in ACT-MI. Because PCT has been established as an evidence-based active control condition, it is likely to serve as a beneficial transdiagnostic intervention in its own right.
  Other Names: PCT-MI
  Arms: Present Centered Therapy for Moral Injury (PCT-MI)

SUMMARY:
The need for moral injury interventions is increasingly being recognized as a domain in Veteran care that must be addressed. Consequences of exposure to morally injurious events include risk for suicide, substance abuse, and refractory symptoms of PTSD and depression. Exposure to morally injurious events is also highly prevalent among Veterans. Thus, interventions addressing moral injury are crucial to helping Veterans build meaningful lives. Psychotherapies explicitly targeting moral injury and functional recovery associated with this construct are limited in VHA. The proposed study serves as a first step in addressing this gap in the literature through the development of a recovery-oriented, evidence-based treatment approach for moral injury among warzone Veterans who report functional impairments related to moral emotions. The proposed pilot study will evaluate the acceptability of this intervention and the feasibility of the design for a future study to test the treatment's capacity to improve patients' functioning.

DETAILED DESCRIPTION:
Warzone Veterans exposed to morally injurious events frequently experience numerous difficulties in functioning. These Veterans often report suicidal ideation and behavior, substance abuse, symptoms of depression and PTSD, and problems in resuming valued living (e.g., spiritual practice, close relationships). Despite the transdiagnostic nature of moral injury, there are no moral injury-specific transdiagnostic interventions. Existing interventions tend to be focused on treating moral injury in the context of PTSD. In addition to an emphasis on PTSD, these interventions target beliefs associated with moral injury as causal factors in the development and maintenance of suffering. An emphasis on altering beliefs associated with moral injury may not optimally facilitate functional recovery as moral pain from moral violations may be justified. As one third of warzone Veterans endorse exposure to morally injurious events, it is vital to develop interventions that can be efficiently disseminated in VHA to facilitate functional recovery. The ideal intervention must simultaneously address moral emotions and promote values consistent behavior in the face of these emotions.

Acceptance and Commitment Therapy for moral injury (ACT-MI) is a recovery-based, psychosocial treatment ideally suited for Veterans endorsing difficulties in functioning related to moral injury. ACT teaches skills to help Veterans relate differently to painful thoughts, emotions, urges, and sensations. Rather than focusing on symptom reduction, ACT is an evidence-based intervention that directly targets functional recovery by assisting Veterans in identifying and engaging in values-consistent behavior even in the presence of distress. In Veteran populations specifically, ACT has been demonstrated effective in treating suicidal ideation and depression and as a result, has been "rolled-out" as an evidence based psychotherapy for depression within VHA. ACT-MI operates on the principles of ACT, with an explicit focus on the social functions of moral emotions. ACT-MI is the only intervention for moral injury that is based on social functionalism which purports that moral emotions (e.g., shame, pride) serve evolutionary purposes essential to group survival. Thus learning to interact with moral emotions differently is crucial to recovery. In ACT-MI, a group-based intervention is used to facilitate in-vivo exposure to moral emotions in the context of values. The proposed two arm randomized controlled pilot study will evaluate the acceptability of ACT-MI and an active control treatment, and determine the feasibility of the randomized controlled trial design for a future full-scale efficacy study. To accomplish this goal the investigators will continue to refine ACT-MI. Veterans enrolled will be randomized to: (a) Present Centered Therapy (PCT) or (b) ACT-MI, both of which will consist of 12, 90-minute group sessions. The specific aims of this study are to: (1) Evaluate the acceptability of the ACT-MI intervention for Veterans experiencing impairment in functioning associated with moral injury, (2) Determine the feasibility of the efficacy study design, and to (3) Select measures and calculate the necessary sample size for a future efficacy study. The performance of validated scales will be measured, in addition to selected NIH Patient Reported Outcomes Measurement Information System modules. All participants will complete a baseline assessment, post treatment, and follow-up assessment one and three months after completion of ACT-MI or PCT. Participants in both groups will also complete a post-treatment assessment on the acceptability of the intervention. The proposed study represents a crucial first step in a line of research likely to yield a recovery oriented, empirically-supported intervention for moral injury among Veterans. The objectives of ACT-MI directly align with Rehabilitation Research and Development's goal to improve Veteran functioning, increase community reintegration, and to facilitate Veteran centered care.

Note, as of March 7, 2024: Completed recruitment for baselines, still collecting data for post treatment, 1-month, and 3-month follow-ups

ELIGIBILITY:
Inclusion Criteria:

* Eligible for VHA care
* Has been deployed to a warzone
* Has experienced a morally injurious event which continues to interfere with functioning
* Willing to be randomized and participate in either of the two conditions

Exclusion Criteria:

* Inability to provide informed consent
* Inability to complete study measures, e.g.:

  * due to significant acute intoxication/withdrawal symptoms
  * mania
  * psychosis
  * aggression
  * catatonia
  * cognitive impairment
* Imminent suicide risk
* Membership in a vulnerable population, e.g.:

  * pregnant women
* History of significant violence towards VA staff
* Participation in another psychotherapy research study
* Current participation in an EBP for a condition related to moral injury

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Borges, PhD, Principal Investigator — Rocky Mountain Regional VA Medical Center, Aurora, CO
Locations (1):
- Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Acceptance and Commitment Therapy for Moral Injury (ACT-MI): Acceptance and Commitment Therapy for Moral Injury (ACT-MI) is a novel treatment protocol detailing the application of ACT for recovery from moral injury. ACT-MI is designed to help Veterans learn to interact differently with moral emotions and engage meaningfully in their lives. The fifteen session intervention is a hybrid group and individual treatment spanning twelve, 90-minute sessions and three 30-minute individual case conceptualization sessions at the beginning, middle, and end of treatment. The current ACT-MI protocol was developed through an iterative process in which authors generated and refined the intervention based on clinical interactions with Veterans currently reporting moral injury. ACT-MI is designed to help Veterans learn to interact differently with moral emotions and engage meaningfully in their lives.
- Present Centered Therapy for Moral Injury (PCT-MI): Present Centered Therapy for Moral Injury (PCT-MI) was adapted from the version of PCT used in PTSD clinical trials (Frost et al., 2014; Wattenberg et al., 2021) to include moral injury psychoeducation and individual case conceptualization sessions consistent with a process-based theoretical framework. PCT-MI is a fifteen session intervention consisting of a hybrid of twelve 90-minute group psychotherapy sessions and three 30-minute individual case conceptualization sessions at the beginning, middle, and end of treatment. PCT-MI group sessions are process-based and emphasize problem-solving moral injury-related life issues.
Period: Pre-Treatment and Randomization
Arm/Group | Acceptance and Commitment Therapy for Moral Injury (ACT-MI) | Present Centered Therapy for Moral Injury (PCT-MI)
Started | 38 | 36
Completed | 37 | 36
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Treatment
Arm/Group | Acceptance and Commitment Therapy for Moral Injury (ACT-MI) | Present Centered Therapy for Moral Injury (PCT-MI)
Started | 37 | 36
Completed | 27 | 21
Not Completed | 10 | 15
Not completed — Attended less than 70% of sessions | 10 | 15
Period: Post-Treatment Assessment
Arm/Group | Acceptance and Commitment Therapy for Moral Injury (ACT-MI) | Present Centered Therapy for Moral Injury (PCT-MI)
Started | 29 | 27
Completed | 29 | 27
Not Completed | 0 | 0
Period: One-Month Follow-Up Assessments
Arm/Group | Acceptance and Commitment Therapy for Moral Injury (ACT-MI) | Present Centered Therapy for Moral Injury (PCT-MI)
Started | 25 | 24
Completed | 25 | 24
Not Completed | 0 | 0
Period: Three-Month Follow-up Assessments
Arm/Group | Acceptance and Commitment Therapy for Moral Injury (ACT-MI) | Present Centered Therapy for Moral Injury (PCT-MI)
Started | 25 | 24
Completed | 25 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acceptance and Commitment Therapy for Moral Injury (ACT-MI) | Present Centered Therapy for Moral Injury (PCT-MI) | Total
Number analyzed (Participants) | 38 | 36 | 74
Age, Continuous [Median (Full Range); unit: years] | 42 [31 to 76] | 40.5 [28 to 72] | 41.5 [28 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 35 | 32 | 67
Race/Ethnicity, Customized [Number; unit: participants]
  White | 28 | 28 | 56
  Black | 1 | 2 | 3
  Native American/Alaskan Native | 1 | 1 | 2
  Asian | 1 | 1 | 2
  Pacific Islander | 2 | 2 | 4
  Multiracial | 3 | 1 | 4
  Other | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38 | 36 | 74
Sexual Orientation [Number; unit: participants]
  Heterosexual | 35 | 32 | 67
  Gay/Lesbian/Queer/Bisexual | 3 | 3 | 6
  Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Client Satisfaction Questionnaire
Description: The investigators will assess the proportion of participants who find ACT-MI acceptable, defined as 70% of participants scoring 24 on the Client Satisfaction Questionnaire (CSQ). The total for the CSQ can range from 8- to 32-points. Higher scores on the CSQ indicate greater treatment acceptability.
Time Frame: Post-treatment (0-7 days after treatment completion)
Population: Post-treatment data were collected from all participants who completed at least one treatment session. 9 participants were lost to follow-up from ACT-MI and 9 participants were lost to follow-up from PCT-MI.
Measure: Count of Participants; unit: Participants
Arm/Group | Acceptance and Commitment Therapy for Moral Injury (ACT-MI) | Present Centered Therapy for Moral Injury (PCT-MI)
Number analyzed (Participants) | 29 | 27
Participants | 27 | 22

2. Primary Outcome: Narrative Evaluation of Intervention Interview
Description: The Narrative Evaluation of Intervention Interview (NEII) will be used to inform any necessary revisions to the intervention and refinement of the treatment manual. The NEII is a semi-structured qualitative interview assessing the perspective of each participant about the impact of the intervention, helpful and unhelpful components, and comparison to other interventions. The NEII will be used to assess acceptability and inform revisions to the treatment manuals. The NEII includes domains related to description of intervention process, description of intervention outcome, evaluation of intervention process, and evaluation of intervention outcome. Data provided reflects the number of participants who provided perspective feedback.
Time Frame: Post-treatment (0-7 days after treatment completion)
Population: Post-treatment data were collected from all participants who completed at least one treatment session. All participants responded related to each NEII domain. 9 participants were lost to follow-up from ACT-MI and 9 participants were lost to follow-up from PCT-MI.
Measure: Count of Participants; unit: Participants
Arm/Group | Acceptance and Commitment Therapy for Moral Injury (ACT-MI) | Present Centered Therapy for Moral Injury (PCT-MI)
Number analyzed (Participants) | 29 | 27
Participants | 29 | 27

3. Primary Outcome: Reasons for Termination (Client and Therapist Versions)
Description: The Reasons for Termination scale is a self-report measure which assesses the impact of common reasons patients terminate therapy. The scale will be used to assess treatment acceptability. Participants who terminate treatment early and their therapists will be asked to independently rate their reasons for termination in 19 domains. Possible total scores on this scale range from 10 to 190-points. Higher scores indicate that the reason for termination had a very great influence on the participant's termination of therapy.
Time Frame: Post-treatment (0-7 days after terminating treatment)
Population: Data reflects those who terminated treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Acceptance and Commitment Therapy for Moral Injury (ACT-MI) | Present Centered Therapy for Moral Injury (PCT-MI)
Number analyzed (Participants) | 38 | 26
Participants | 10 | 14

4. Secondary Outcome: Valued Living Questionnaire
Description: The Valued Living Questionnaire is a self-report measure that assesses participants' values as well as the consistency with which they believe they have been living life according to their values. This scale will be examined as a candidate outcome measure for a future efficacy trial. A possible of 10 to 100 total points for importance of values and 10 to 100 total points for consistency of action with values is demonstrated on the Valued Living Questionnaire (VLQ). Higher scores on the VLQ are indicative of greater importance of values and greater consistency in acting on values.
Time Frame: Pre-treatment (Up to 30-days before starting treatment), post-treatment (0-7 days after treatment completion) and 1- and 3-month follow-up
Population: The number of participants analyzed in row two and three differ from row one because the results are from different time points and some participants were lost to follow up.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Acceptance and Commitment Therapy for Moral Injury (ACT-MI) | Present Centered Therapy for Moral Injury (PCT-MI)
Number analyzed (Participants) | 37 | 36
score on a scale
  Pre-Treatment | 40.9 [35.06 to 46.74] | 41.55 [36.12 to 46.98]
  Post-Treatment: number analyzed (Participants) | 29 | 27
  Post-Treatment | 49.83 [42.95 to 56.73] | 42.63 [35.88 to 49.99]
  One-Month Follow-Up: number analyzed (Participants) | 25 | 24
  One-Month Follow-Up | 50.16 [42.01 to 58.31] | 42.01 [34.69 to 49.33]
  Three-Month Follow-Up: number analyzed (Participants) | 25 | 23
  Three-Month Follow-Up | 45.77 [38.15 to 53.39] | 41.82 [35.55 to 48.09]

5. Secondary Outcome: Outcome Questionnaire-45 (OQ-45)
Description: The Outcome Questionnaire-45 (OQ-45) is a self-report measure that assesses functioning in the psychosocial domains of symptom distress (0-100 points), social relations (0-44 points), and social role functioning (0-36 points). The OQ-45 will be examined as a candidate outcome measure for a future efficacy trial. Higher scores on the OQ-45 are indicative of more symptom distress, difficulty in social relations, and difficulty in social role functioning.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Acceptance and Commitment Therapy for Moral Injury (ACT-MI) | Present Centered Therapy for Moral Injury (PCT-MI)
Number analyzed (Participants) | 37 | 36
score on a scale
  Pre-Treatment | 69.89 [64 to 75.78] | 69.78 [63.11 to 76.45]
  Post-Treatment: number analyzed (Participants) | 29 | 27
  Post-Treatment | 53.62 [45.22 to 62.02] | 63.30 [59.79 to 78.81]
  One-Month Follow-Up: number analyzed (Participants) | 25 | 24
  One-Month Follow-Up | 60.76 [51.34 to 70.18] | 66.92 [57.69 to 76.15]
  Three-Month Follow-Up: number analyzed (Participants) | 25 | 24
  Three-Month Follow-Up | 63.76 [54.07 to 73.45] | 63.21 [53.37 to 73.05]

6. Secondary Outcome: PROMIS Short Form v2.0-Satisfaction With Social Roles and Activities 8a
Description: This is a self-report measure that assesses ability to perform various social activities. This measure will be examined as a candidate outcome measure for a future efficacy trial. Total scores range from 8 to 40 points on this scale with higher scores associated with greater satisfaction with social roles and activities.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Acceptance and Commitment Therapy for Moral Injury (ACT-MI) | Present Centered Therapy for Moral Injury (PCT-MI)
Number analyzed (Participants) | 36 | 36
score on a scale
  Pre-Treatment | 21.53 [18.84 to 24.22] | 21.33 [18.84 to 23.82]
  Post-Treatment: number analyzed (Participants) | 29 | 27
  Post-Treatment | 27.14 [24.23 to 30.05] | 25.33 [21.79 to 28.87]
  One-Month Follow-Up: number analyzed (Participants) | 25 | 25
  One-Month Follow-Up | 24.92 [21.89 to 27.95] | 23.28 [20.39 to 26.17]
  Three-Month Follow-Up: number analyzed (Participants) | 24 | 23
  Three-Month Follow-Up | 23.96 [20.16 to 27.76] | 23.91 [20.90 to 26.92]

7. Secondary Outcome: PROMIS v2.0-Social Isolation
Description: This is a self-report measure that assesses experience of social isolation. This measure will be examined as a candidate outcome measure for a future efficacy trial. Total scores range from 4 to 20 points with higher scores on this scale associated with greater social isolation.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Acceptance and Commitment Therapy for Moral Injury (ACT-MI) | Present Centered Therapy for Moral Injury (PCT-MI)
Number analyzed (Participants) | 37 | 36
score on a scale
  Pre-Treatment | 14.14 [12.90 to 15.38] | 14.39 [13.36 to 15.42]
  Post-Treatment: number analyzed (Participants) | 29 | 27
  Post-Treatment | 12.24 [10.80 to 13.68] | 13.22 [11.79 to 14.65]
  One-Month Follow-Up: number analyzed (Participants) | 25 | 25
  One-Month Follow-Up | 13.40 [11.83 to 14.97] | 14.08 [12.72 to 15.42]
  Three-Month Follow-Up: number analyzed (Participants) | 25 | 23
  Three-Month Follow-Up | 13.48 [11.92 to 15.04] | 13.78 [11.94 to 15.62]

8. Secondary Outcome: Ecological Momentary Assessment
Description: Self-report ecological momentary assessment via a smart phone application was developed to assess in the moment experiential avoidance, emotions, and engagement in valued behavior. However, because VA regulations and use of a new application, analyses will focus on feasibility of completing the EMA and will be reported as number of participants who provided EMA data. Actual EMA responses will only be analyzed if there is sufficient participation. Actual EMA responses will only be analyzed if there are 25% or more reporting participants.
Time Frame: Pre-treatment (Up to 30-days before starting treatment for a 1-week period) and post-treatment (0-7 days after treatment completion for a 1-week period)
Population: EMA procedures tested proved not to be feasible and resulted in a problematic amount of missing data. Most Veterans chose not to participate largely due to the need to present to the VA in person to return the data due to VA regulatory barriers.
Measure: Count of Participants; unit: Participants
Arm/Group | Acceptance and Commitment Therapy for Moral Injury (ACT-MI) | Present Centered Therapy for Moral Injury (PCT-MI)
Number analyzed (Participants) | 38 | 36
Participants | 9 | 5

9. Secondary Outcome: Inventory of Psychosocial Functioning
Description: Self-report measure that assesses impairment within the last 30 days across a spectrum of psychosocial domains. Will be examined as a candidate outcome measure for a future efficacy trial. Response options range from 0 = never to 6 = always. The measure yields a mean score for the total scale. Higher scores indicate less functional impairment. The total scale score is reported.
Time Frame: Pre-treatment, post-treatment, one-month follow-up, and three-month follow-up
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Acceptance and Commitment Therapy for Moral Injury (ACT-MI) | Present Centered Therapy for Moral Injury (PCT-MI)
Number analyzed (Participants) | 37 | 36
score on a scale
  Pre-Treatment | 2.78 [2.56 to 3] | 2.77 [2.58 to 2.96]
  Post-Treatment: number analyzed (Participants) | 29 | 27
  Post-Treatment | 2.41 [2.17 to 2.65] | 2.57 [2.33 to 2.81]
  One-Month Follow-Up: number analyzed (Participants) | 25 | 25
  One-Month Follow-Up | 2.43 [2.14 to 2.72] | 2.74 [2.40 to 3.08]
  Three-Month Follow-Up: number analyzed (Participants) | 25 | 23
  Three-Month Follow-Up | 2.51 [2.21 to 2.81] | 2.64 [2.39 to 2.89]

ADVERSE EVENTS:
Time Frame: Data were collected from August of 2019 to October of 2024. Each participant was active in the study (treatment sessions and assessment sessions) for approximately 8 months.
Arm/Group | Acceptance and Commitment Therapy for Moral Injury (ACT-MI) | Present Centered Therapy for Moral Injury (PCT-MI)
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/36
Other Adverse Events (participants affected / at risk) | 0/38 | 0/36

LIMITATIONS AND CAVEATS:
Outcome data are provided, but should not be used to draw conclusions about the efficacy of ACT-MI given recommendations for pilot study best practices (e.g., Eldridge et al., 2016) and data lost to follow up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-01-17): https://cdn.clinicaltrials.gov/large-docs/31/NCT03760731/Prot_SAP_ICF_000.pdf